CLINICAL TRIAL: NCT02488954
Title: Interest of Propionibacterium Freudenreichii for the Treatment of Mild to Moderate Ulcerative Colitis
Acronym: EMMENTAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-000835-34; 35RC14_9817_EMMENTAL (Other: CHU de Rennes)
Record Dates: First submitted 2015-06-23; First posted 2015-07-02 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Probiotics; treatments; Propionibacterium freudenreichii
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics (Experimental): Oral daily take of probiotics in the form of cheese portion (50g) during 8 weeks
  Interventions: Other: Probiotics in the form of cheese portion

INTERVENTIONS:
Other: Probiotics in the form of cheese portion

SUMMARY:
Ulcerative colitis (UC) is an immune mediated chronic inflammatory bowel disease that results at least in part of an abnormal immune response to environmental factors including the intestinal microbiota. Thus, use of probiotics (microorganisms that are believed to provide health benefits when consume) may restore the gastrointestinal microbiota and reduce intestinal inflammation.

Propionibacterium freudenreichii is used for the production of fermented food products (cheese). Some selected strains have strong anti-inflammatory properties. Use of cheese based on a monoxenic culture of anti-inflammatory strain of Propionibacterium freudenreichii may decrease disease activity during ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age above 18 years old
* Patient with diagnosis of ulcerative colitis for at least 6 months.
* Patient with mayo endoscopic score ≥ 1
* Patient with mild to moderate disease activity (3 < SCCI < 12)
* Ongoing treatment by mesalamine, steroids, thiopurines or Tumor Necrosis Factor antagonist at stable dose.
* Patients who have given written informed consent.

Exclusion Criteria:

* Adults legally protected (under judicial protection, guardianship, or supervision), persons deprived of their liberty.
* Psychiatric disease that alter the judgment
* Stoma
* Proctocolectomy
* Severe disease (SCCI >12, acute severe colitis)
* Steroid dose > 10 mg/j or introduction of steroid (topic or oral) within 4 weeks
* Introduction or dose optimization of TNF antagonist within 4 months
* Introduction or dose optimization of thiopurine
* Hemoglobin level < 11,5 g/dL, Platelets > 400000/mm3, Leukocytosis > 10 000/mm3
* Intolerant to lactose
* Disease extent limited to the rectum
* Mayo endoscopic subscore of 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Response rate | Week 8
  Response rate is defined by a decrease of at least two points of the Simple Clinical Colitis Index (SCCI)

SECONDARY OUTCOMES:
Rate of clinical response | Week 4
Rate of clinical remission | Week 4
  Clinical remission rate is defined by a SCCI<3
Rate of clinical remission | Week 8
  Clinical remission rate is defined by a SCCI<3
Rate of mucosal healing | Week 8
  Mucosal Healing is defined by a Mayo endoscopic subscore of 0 or 1
Rate of deep (clinical and endoscopic) remission | Week 8
  Deep remission is defined clinically and by endoscopic exams
Side effects | Week 8
  Assessment of adverse events
Rate of response based on presence of Proprionibacterium freudenreichii in stools at week 0 | Week 8
  Proprionibacterium freudenreichii analysis in stools
Remission rate based on presence of Proprionibacterium freudenreichii in stools at week 0 | Week 8
  Proprionibacterium freudenreichii analysis in stools

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France